CLINICAL TRIAL: NCT00724880
Title: Effect of Clopidogrel (Plavix) on Postoperative Bleeding in Patients Undergoing Coronary Artery Bypass Surgery. A Prospective Randomized Controlled Study
Brief Title: Effect of Clopidogrel (Plavix) on Postoperative Bleeding in Patients Undergoing Coronary Artery Bypass Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Drs. Firanescu, Catharina hospital, department of cardiothoracic surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Plavix studie
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass grafting; clopidogrel; post-operative bleeding
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

ARMS (3):
- 1 (Experimental): Clopidogrel is stopped 5 days prior to surgery
  Interventions: Drug: Clopidogrel
- 2 (Experimental): Clopidogrel is stopped 3 days prior to surgery
  Interventions: Drug: Clopidogrel
- 3 (Experimental): Clopidogrel is stopped 0 days prior to surgery
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel is stopped 5 days prior to surgery
  Other Names: plavix
  Arms: 1
Drug: Clopidogrel — Clopidogrel is stopped 3 days prior to surgery
  Other Names: plavix
  Arms: 2
Drug: Clopidogrel — Clopidogrel is stopped 0 days prior to surgery
  Other Names: plavix
  Arms: 3

SUMMARY:
* Running title: Effect of Clopidogrel on Postoperative Bleeding in Patients undergoing Coronary Artery Bypass Surgery
* Title: Clopidogrel and bleeding in patients undergoing coronary artery bypass grafting. Is surgical delay necessary in patients using clopidogrel? And if so, which is the safety time interval when clopidogrel should be stopped before surgery in order to avoid bleeding and other related complications.
* Background: By blockade of the platelet ADP receptor, clopidogrel inhibits the binding of fibrinogen to the platelet GPIIb/IIIa receptor complex, thereby preventing platelet aggregation from ADP stimulation. Some authors suggest that the platelet function is completely recovered in 7 days after stopping clopidogrel in healthy subjects. Other researches suggest full recovery of platelet function in 3 to 5 days.
* Study objectives: To investigate if the interruption of the clopidogrel is necessary before CABG in order to prevent bleeding and other complications.

To trace the increased risk patients for postoperative bleeding and to individualize the therapy according to TEG measurements.

* Design: A prospective, randomized mono- center study
* Patients: Patients who are receiving elective or urgent CABG surgery and are pre-treated at least 5 days before surgery with clopidogrel
* Primary endpoint: To determine if there are significant differences in blood loss, transfusions and rethoracotomies in the three selected groups of patients treated with clopidogrel To asses the predictive value of the TEG clot strength in postoperative bleeding in patients using Clopidogrel.
* Secondary endpoints: Death, myocardial infarction, stroke, respiratory failure, renal failure requiring dialysis, mediastinitis,readmission rates within 30 days from discharge, and ICU and hospital lengths of stay
* Risks: Using standard dose of aprotinin, we consider no increased risk in blood loss and other related complications for this three groups of patients.
* Possible benefits: Reduction of time delay in operating patients under treatment with clopidogrel.

A more accurate time interval when clopidogrel should be stopped before surgery in order to eliminate the risk of bleeding and associated complications.

ELIGIBILITY:
Inclusion criteria:

1. Patients who are using clopidogrel at least 5 days before surgery with a dose of 75 mg clopidogrel without loading dose with or without concomitant use of aspirin.
2. Patients who received a loading dose of 300-600 mg clopidogrel 24 hours before CABG, with or without concomitant use of aspirin
3. Patients approved for elective or urgent CABG surgery

Exclusion criteria:

1. Patients who are concomitant using oral coumarin derivates, heparine derivates iv., dipiridamol or other anticoagulant treatment, 5 days before operation.
2. Patients with pre-existing bleeding disorders, thrombocytopenia
3. Patients who have renal insufficiency (creatinine >2.0 mg/dL) or chronic renal failure requiring dialysis
4. Patients in end stage heart failure
5. Patients who have evidence of significant hepatic disease including clinical signs or laboratory values of total bilirubin> 2.0 mg/dL, ALAT or ASAT> 3X upper limit of normal, or INR >2X upper limit of normal (not due to anticoagulation therapy)
6. Emergency bypass surgery when patients cant be random enrolled in one of the three groups
7. Concomitant valvular or other cardiac procedures
8. Re-operation (patients known with previous heart operations)
9. Off-pump CABG
10. Chronic alcoholism
11. Immediate post operative complications that in the opinion of the investigator can alter the further results of the trial (thromboembolism or ischemic CVA with use of anticoagulants, severe liver function disorders, sepsis, disseminated intravascular coagulation, adverse effects to blood products, etc)
12. Patients whom recently (3-6 months before screening) received PCI and continuation of clopidogrel till the day of operation is advisable (according to the advice of the cardiologist)
13. Patients who refuse to accept medically- indicated blood products
14. Pregnancy and breast feeding
15. Patients who received investigational drugs in the previous 30 days, or are currently participating in a study during which the administration of investigational drugs within one month is anticipated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary end point of this study is to determine if there are significant differences in blood loss, transfusions and rethoracotomies in the three selected groups of patients treated with clopidogrel | within 30 days (+/- 5 days) after surgery
To asses the predictive value of the TEG clot strength in postoperative bleeding in patients using clopidogrel | within 30 days (+/- 5 days) after surgery

SECONDARY OUTCOMES:
death | within 30 days (+/- 5 days) after surgery
myocardial infarction | within 30 days (+/- 5 days) after surgery
stroke | within 30 days (+/- 5 days) after surgery
respiratory failure | within 30 days (+/- 5 days) after surgery
renal failure requiring dialysis | within 30 days (+/- 5 days) after surgery
mediastinitis | within 30 days (+/- 5 days) after surgery
wound infection | within 30 days (+/- 5 days) after surgery
readmission rates within 30 days from discharge | within 30 days (+/- 5 days) after surgery
ICU and hospital lengths of stay. | within 30 days (+/- 5 days) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: A.H.M. van Straten, MD, Principal Investigator — Catharina hospital, department of Cardio Thoracic Surgery